CLINICAL TRIAL: NCT00852163
Title: Phase II Trial of Clofarabine With Parenteral Busulfan (Busulfex®) Followed by Allogeneic Related or Unrelated Donor Transplantation for the Treatment of Hematologic Malignancies and Diseases
Brief Title: Study of Stem Cell Transplant for Leukemia and Myelodysplastic Syndromes Using Clofarabine and Busulfan Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 006-150
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia; Myelodysplastic Syndrome
Keywords: conditioning, preparative; clofarabine; transplant; Busulfan; leukemia; myelodysplastic syndrome
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Clofarabine; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine with Busulfan (Experimental): Clofarabine 40 mg/m2 IV QD × 5 days Busulfan (Busulfex™) 3.2 mg/kg IV QD × 2 days
  Interventions: Drug: Clofarabine with Busulfan

INTERVENTIONS:
Drug: Clofarabine with Busulfan — Clofarabine 40 mg/m2 IV QD × 5 days Busulfan (Busulfex™) 3.2 mg/kg IV QD × 2 days
  Other Names: Clofarabine:CLOLAR, clofarabine; CAFdA; Cl-F-ara-A;; Busulfan: Busulfex™

SUMMARY:
The purpose of this study is to determine whether Clofarabine in combination with Busulfan is effective as a preparative transplant regimen for the treatment of leukemia and myelodysplastic syndromes

DETAILED DESCRIPTION:
The success of allogeneic hematopoietic transplantation in the treatment of myeloid malignancies is determined by two main factors: the limiting of regimen-related toxicity and the prevention of recurrent leukemia. Over the past 10 years, considerable clinical research has been devoted to the reduction of regimen-related toxicity through the use of reduced-intensity (nonmyeloablative) transplants. However, leukemic relapse has remained a difficult obstacle. Thus, the need for highly effective, yet non-toxic regimens persists, particularly for elderly patients for whom very little overall progress has been made. Clofarabine is a chemotherapeutic agent with novel myelotoxic properties and proven low toxicity in older patients. These qualities suggest clofarabine may be a useful component of conditioning regimens for stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

Disease Criteria:

* Acute myelogenous leukemia (AML)
* Acute lymphocytic leukemia (ALL)
* Myelodysplastic syndromes (MDS) Refractory anemia (RA) with adverse cytogenetics (SWOG criteria) or beyond (RAEB, RAEB-T, AML)
* Other Myeloproliferative Disorders Myelofibrosis, Agnogenic Myeloid Metaplasia, Chronic Myelomonocytic Leukemia (CMML)
* Chronic lymphocytic leukemia (CLL) High risk or advanced disease

Other Inclusion Criteria:

* 18 years of age or older
* Related or unrelated donor with HLA criteria as follows:

  * Related donors: a serologic equivalent HLA Class I (A, B, and C) and Class II DRB1 or DQB1 matched donor OR a donor who is a single 1 antigen mismatched for A, B, C, DRB1, or DQB1 loci
  * Unrelated donors: sequence-based typing fully matched A, B, C, DRB1, and DQB1 allele-matched donor OR a donor who is no greater than 1 antigen mismatched for A, B, C, DRB1, or DQB1 loci
* Able to provide valid informed consent.
* Female patients must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for up to 12 months after study treatment.

Exclusion Criteria:

Organ Function Criteria:

* Cardiac: symptomatic coronary artery disease or ejection fraction <45% or uncontrolled cardiac failure
* Pulmonary: FEV1 or DLCO (corrected) <50% of predicted values and/or receiving continuous supplementary oxygen
* Hepatic: Bilirubin ≥ 1.2 mg/dL or AST/ALT ≥ 3x upper limit of normal (ULN) unless the liver is involved with malignant disease
* Renal: creatinine clearance < 60 mL/min (24-hour urine collection) or <50 mL/min (Glofil test)
* Karnofsky score <60%
* Active CNS disease
* Prior hematopoietic transplantation (autologous or allogeneic) <6 months prior to study entry
* Use of investigational agents less than or equal to 30 days before study entry.
* Life threatening, or clinically significant infection
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Female patients who are pregnant or breast feeding
* HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-03; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Disease free survival at one and two year | At 1 year and 2 Year

SECONDARY OUTCOMES:
Incidence of hematopoietic engraftment | 100 days
Incidence and severity of acute toxicities | 100 days
Pharmacokinetic profiles of high dose busulfan and standard dose clofarabine | Lesss than 8 days
Acute GVHD | 100 Days

CONTACTS AND LOCATIONS:
Overall Officials: Edward Agura, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States